CLINICAL TRIAL: NCT02559297
Title: Effects of Sevoflurane and Desflurane Anesthesia on Regulatory T Cells in Patients Undergoing Living Donor Kidney Transplantation
Brief Title: Effects of Sevoflurane and Desflurane on Treg
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Arpa Chutipongtanate, Faculty Member, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 04-58-23
Record Dates: First submitted 2015-09-22; First posted 2015-09-24 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Transplant; Failure, Kidney
Keywords: Regulatory T cells; Sevoflurane; Desflurane; Cytokines; Flow cytometry; Living Donor Kidney Transplant
MeSH Terms: interventions — Sevoflurane; Desflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sevoflurane (Active Comparator): In sevoflurane arm (n=20) at the beginning after successful intubation, 2 L/min nitric oxide (N2O), 2 L/min O2 , and 2% to 2.5% sevoflurane will be given for 10 minutes then total flow will be decreased to 2 L/min. Anesthesia will be maintained using 1-1.5 minimal alveolar concentration (MAC) of sevoflurane in 50% O2 and 50% N2O.
  Interventions: Drug: Sevoflurane
- Desflurane (Experimental): In desflurane arm (n=20) at the beginning after successful intubation, 2 L/min N2O, 2 L/min O2, and 6% to 8% desflurane will be given for 10 minutes then total flow will be decreased to 2 L/min. Anesthesia will be maintained using 1-1.5 MAC of desflurane in 50% O2 and 50% N2O.
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Sevoflurane — After induction of anesthesia and successful intubation, 2 L/min N2O, 2 L/min O2 , and 2% to 2.5% sevoflurane will be given for 10 minutes then total flow will be decreased to 2 L/min. Anesthesia will be maintained using 1-1.5 minimal alveolar concentration (MAC) of sevoflurane in 50% O2 and 50% N2O. Ventilation will be adjusted to keep end-tidal carbon dioxide 30-35 mmHg (Tidal volume 7-10 mL/kg).
  Other Names: Ultane
  Arms: Sevoflurane
Drug: Desflurane — After induction of anesthesia and successful intubation, 2 L/min N2O, 2 L/min O2 , and 6% to 8% desflurane will be given for 10 minutes then total flow will be decreased to 2 L/min. Anesthesia will be maintained using 1-1.5 minimal alveolar concentration (MAC) of desflurane in 50% O2 and 50% N2O. Ventilation will be adjusted to keep end-tidal carbon dioxide 30-35 mmHg (Tidal volume 7-10 mL/kg).
  Other Names: Suprane
  Arms: Desflurane

SUMMARY:
This prospective interventional study aims to compare sevoflurane and desflurane anesthetic agents on regulatory T cell (Treg) numbers and its cytokine production in patients undergoing Living Donor Kidney Transplant (LDKT).

DETAILED DESCRIPTION:
All patients with end stage renal disease (ESRD) need renal replacement therapy, either dialysis or kidney transplantation. Dialysis, despite its effectiveness in prolonging ESRD patients' lives, is a burden. Successfulness in kidney transplantation will restore good quality of life in ESRD patients. However, one of the most important complications that lead to transplant failure is graft rejection. It is already known that the pathophysiology of the rejection is immune response. Recent evidence showed that regulatory T cell (Treg) plays a central role in preventing graft rejection by inhibiting recipient alloimmune response (1-3). Characterization of Treg numbers and/or functional changes under various conditions may lead to a new preventive measure and/or a novel therapeutic strategy for graft rejection.

Kidney transplantation is conducted under general anesthesia. Interestingly, several agents used in general anesthesia have also modulated immune functions (4-12). Although the effect of inhalation anesthetic agents on leukocyte count has been shown, the effect on Treg function has totally been unknown. Knowing the effects of inhalation agents on Treg numbers and functions will be beneficial to intraoperative management during transplant surgery, aiming toward reducing the risk of graft rejection in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving 1st living donor kidney transplantation

Exclusion Criteria:

* Hyperacute graft rejection
* Pre-existing autoimmune or immunodeficiency diseases in recipients
* Receiving blood product during 24-h perioperative period
* Patient refuse to participate this study at any time point

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-08-10 (Actual); Primary Completion 2017-06-03 (Actual); Study Completion 2017-06-03 (Actual)

PRIMARY OUTCOMES:
Number of regulatory T cells | Within 24-h peri-operative period
  Assessing change of Treg numbers by flow cytometry from baseline (before exposure to sevoflurane or desflurane) to after exposure to sevoflurane or desflurane for 2-h and 24-h

SECONDARY OUTCOMES:
T lymphocyte cytokine production | Within 24-h peri-operative period
  Assessing change of T lymphocyte cytokine production using Multiplex immunoassay of interleukin (IL)-10, Tumor Necrosis Factor (TGF)-beta, IL-2, Interferon (IFN)-gamma, IL-4, IL-5, IL-13, from baseline (before exposure to sevoflurane or desflurane) to after exposure to sevoflurane or desflurane for 2-h and 24-h

CONTACTS AND LOCATIONS:
Overall Officials: Arpa Chutipongtanate, MD, Principal Investigator — Department of Anesthesia, Faculty of Medicine Ramathibodi Hospital, Mahidol University, Thailand
Locations (1):
- Ramathibodi Hospital, Ratchathewi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Data is obtained by flow cytometry and multiplex immunoassay. The data includes percentages of regulatory T cells and the measured cytokines. The data will be available in the end of study period, 05/2017.

REFERENCES:
- [Background] Edozie FC, Nova-Lamperti EA, Povoleri GA, Scotta C, John S, Lombardi G, Afzali B. Regulatory T-cell therapy in the induction of transplant tolerance: the issue of subpopulations. Transplantation. 2014 Aug 27;98(4):370-9. doi: 10.1097/TP.0000000000000243. PMID 24933458
- [Background] San Segundo D, Millan O, Munoz-Cacho P, Boix F, Paz-Artal E, Talayero P, Morales JM, Muro M, De Cos MA, Guirado L, Llorente S, Pascual J, Arias M, Brunet M, Lopez-Hoyos M. High proportion of pretransplantation activated regulatory T cells (CD4+CD25highCD62L+CD45RO+) predicts acute rejection in kidney transplantation: results of a multicenter study. Transplantation. 2014 Dec 15;98(11):1213-8. doi: 10.1097/TP.0000000000000202. PMID 25083613
- [Background] Lopez-Hoyos M, Segundo DS, Fernandez-Fresnedo G, Marin MJ, Gonzalez-Martin V, Arias M. Regulatory T cells in renal transplantation and modulation by immunosuppression. Transplantation. 2009 Aug 15;88(3 Suppl):S31-9. doi: 10.1097/TP.0b013e3181af7b99. PMID 19667959
- [Background] Zhang T, Fan Y, Liu K, Wang Y. Effects of different general anaesthetic techniques on immune responses in patients undergoing surgery for tongue cancer. Anaesth Intensive Care. 2014 Mar;42(2):220-7. doi: 10.1177/0310057X1404200209. PMID 24580388
- [Background] Schneemilch CE, Hachenberg T, Ansorge S, Ittenson A, Bank U. Effects of different anaesthetic agents on immune cell function in vitro. Eur J Anaesthesiol. 2005 Aug;22(8):616-23. doi: 10.1017/s0265021505001031. PMID 16119599
- [Background] Ji FH, Wang YL, Yang JP. Effects of propofol anesthesia and sevoflurane anesthesia on the differentiation of human T-helper cells during surgery. Chin Med J (Engl). 2011 Feb;124(4):525-9. PMID 21362275
- [Background] Pirbudak Cocelli L, Ugur MG, Karadasli H. Comparison of effects of low-flow sevoflurane and desflurane anesthesia on neutrophil and T-cell populations. Curr Ther Res Clin Exp. 2012 Feb;73(1-2):41-51. doi: 10.1016/j.curtheres.2012.02.005. PMID 24653511
- [Background] Loop T, Dovi-Akue D, Frick M, Roesslein M, Egger L, Humar M, Hoetzel A, Schmidt R, Borner C, Pahl HL, Geiger KK, Pannen BH. Volatile anesthetics induce caspase-dependent, mitochondria-mediated apoptosis in human T lymphocytes in vitro. Anesthesiology. 2005 Jun;102(6):1147-57. doi: 10.1097/00000542-200506000-00014. PMID 15915027
- [Background] Hisano T, Namba T, Hashiguchi-Ikeda M, Ito T, Hirota K, Fukuda K. Inhibition of E-selectin-mediated leukocyte adhesion by volatile anesthetics in a static condition. J Anesth. 2005;19(1):1-6. doi: 10.1007/s00540-004-0274-0. PMID 15674507
- [Background] Koksoy S, Sahin Z, Karsli B. Comparison of the effects of desflurane and bupivacaine on Th1 and Th2 responses. Clin Lab. 2013;59(11-12):1215-20. doi: 10.7754/clin.lab.2013.120413. PMID 24409654
- [Background] Kim WH, Jin HS, Ko JS, Hahm TS, Lee SM, Cho HS, Kim MH. The effect of anesthetic techniques on neutrophil-to-lymphocyte ratio after laparoscopy-assisted vaginal hysterectomy. Acta Anaesthesiol Taiwan. 2011 Sep;49(3):83-7. doi: 10.1016/j.aat.2011.08.004. Epub 2011 Sep 22. PMID 21982167
- [Background] Zhou D, Gu FM, Gao Q, Li QL, Zhou J, Miao CH. Effects of anesthetic methods on preserving anti-tumor T-helper polarization following hepatectomy. World J Gastroenterol. 2012 Jun 28;18(24):3089-98. doi: 10.3748/wjg.v18.i24.3089. PMID 22791944
- [Derived] Chutipongtanate A, Prukviwat S, Pongsakul N, Srisala S, Kamanee N, Arpornsujaritkun N, Gesprasert G, Apiwattanakul N, Hongeng S, Ittichaikulthol W, Sumethkul V, Chutipongtanate S. Effects of Desflurane and Sevoflurane anesthesia on regulatory T cells in patients undergoing living donor kidney transplantation: a randomized intervention trial. BMC Anesthesiol. 2020 Aug 27;20(1):215. doi: 10.1186/s12871-020-01130-7. PMID 32854613